CLINICAL TRIAL: NCT04849715
Title: A Phase 3, Randomized, Double-Blind Study Comparing Parsaclisib, a PI3Kδ Inhibitor, in Combination With Bendamustine and Rituximab (BR), With Placebo and BR for the Treatment of Newly Diagnosed Mantle Cell Lymphoma
Brief Title: A Study of Parsaclisib, a PI3Kδ Inhibitor, in Combination With Bendamustine and Rituximab in Patients With Newly Diagnosed Mantle Cell Lymphoma
Acronym: CITADEL-310
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: business decision; no enrolled patients
Sponsor: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: INCB 50465-310
Record Dates: First submitted 2021-04-16; First posted 2021-04-19 (Actual); Last update posted 2022-04-29 (Actual); Status verified 2022-04

CONDITIONS: Mantle Cell Lymphoma
Keywords: parsaclisib; newly diagnosed; bendamuastine; rituximab; PI3Kδ
MeSH Terms: conditions — Lymphoma, Mantle-Cell | interventions — parsaclisib; Rituximab; Bendamustine Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Treatment Group A (Active Comparator): Participants will be administered parsaclisib once daily and will receive Bendamustine and Rituximab periodically for 6 months.
  Interventions: Drug: parsaclisib; Drug: rituximab; Drug: bendamustine
- Treatment group B (Placebo Comparator): Participants will be administered placebo once daily and will receive Bendamustine and Rituximab periodically for 6 months.
  Interventions: Drug: rituximab; Drug: bendamustine; Drug: Placebo

INTERVENTIONS:
Drug: parsaclisib — parsaclisib will be administered orally once daily.
  Other Names: INCB050465
  Arms: Treatment Group A
Drug: rituximab — rituximab is administered IV on Day 1 of each 28-day cycle for 6 cycles.
  Other Names: Rituxan
Drug: bendamustine — bendamustine is administered IV on Day 1 and 2 of each 28-day cycle for 6 cycles.
  Other Names: Bendeka; Treanda
Drug: Placebo — placebo will be administered orally once daily
  Arms: Treatment group B

SUMMARY:
This is a Phase 3, double-blind, randomized, placebo-controlled, multicenter study of parsaclisib plus BR versus placebo plus BR as first-line treatment of participants with newly diagnosed MCL.

ELIGIBILITY:
Inclusion Criteria:

* Male and female participants aged 18 years or older. (Japan aged 20 years or older.)
* Have received no previous systemic anti-lymphoma therapies.
* Pathologically confirmed MCL by local laboratory.
* Histologically confirmed CD20 expression (by flow cytometry or immunohistochemistry) of the MCL cells as assessed by pathology.
* Ineligible for high-dose chemotherapy and autologous stem cell transplantation.
* Radiographically (CT, MRI) measurable lymphadenopathy per the Lugano criteria for response assessment (Cheson et al 2014).
* ECOG PS of 0 to 2.
* Willingness to avoid pregnancy or fathering children.

Exclusion Criteria:

* Presence of any lymphoma other than MCL.
* Presence of CNS lymphoma (either primary or secondary) or leptomeningeal disease.
* Requires treatment with potent inducers and inhibitors of CYP3A4
* Inadequate organ functions including hematopoiesis, liver, and kidney significant concurrent, uncontrolled medical condition, including, but not limited to, renal, hepatic, hematological, GI, endocrine, pulmonary, neurological, cerebral, or psychiatric disease.
* History of other malignancy within 2 years of study entry.
* Known HIV infection, HBV or HCV.
* HBV or HCV infection: Participants positive for HBsAg or anti-HBc will be eligible if they are negative for HBV-DNA; these participants must receive prophylactic antiviral therapy. Participant's positive for HCV antibody will be eligible if they are negative for HCV-RNA.
* Clinically significant cardiac disease, congestive heart failure, including unstable angina, acute myocardial infarction, or cardiac conduction issues, within 6 months of randomization.
* Abnormal ECG findings that are clinically meaningful per investigator's assessment.
* Women who are pregnant or breastfeeding
* Any condition that would, in the investigator's judgment, interfere with full participation in the study, including administration of study treatment and attending required study visits; pose a significant risk to the participant; or interfere with interpretation of study data.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-03-11 (Estimated); Primary Completion 2030-08-15 (Estimated); Study Completion 2034-07-07 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival | 7 years
  Defined as the time from the date of randomization until the date of first-documented disease progression, as determined by an Independent Review Committee (IRC) based on the Lugano criteria, or death from any cause, whichever happens first.

SECONDARY OUTCOMES:
Overall Survival | 10 years
  Defined as the time from the date of randomization until death from any cause.
Objective Response Rate | 7 Years
  Defined as the proportion of participants with a Complete Response (CR) or Partial Response (PR) as determined by an IRC- provided radiographic disease assessment of response according to response criteria for lymphomas.
Complete Response Rate | 7 Years
  Defined as the proportion of participants with a CR as determined by an IRC- provided radiographic disease assessment of response according to response criteria for lymphomas.
Duration of Response | 7 Years
  Defined as the time from first-documented evidence of CR or PR until first documented disease progression or death from any cause, whichever happens first, among participants who achieve an objective response, as determined by radiographic disease assessment provided by an IRC.
Duration Of Complete Response | 7 Years
  Defined as the time from the first evidence of CR to the date of first documented disease progression or death from any cause, whichever happens first, among participants who achieve a CR, as determined by radiographic disease assessment provided by an IRC.
Disease Control Rate | 7 Years
  Defined as the proportion of participants who achieved a response of CR, PR, or Stable Disease (SD) assessed by an IRC.
Event Free Survival | 7 Years
  Defined as the time from date of randomization to date of first documented progression, as determined by radiographic disease assessment provided by an IRC, administration of a new anti lymphoma treatment, or death from any cause, whichever happens first.
Time To Next anti-Lymphoma Treatment | 7 Years
  Defined as the time from date of randomization to date of first documented administration of a new anti-lymphoma treatment.
Progression-Free Survival on next anti-lymphoma treatment | 7 Years
  Defined as the time from the date of randomization to the date of first documented disease progression as reported by investigator after next anti-lymphoma treatment or death from any cause, or start of a third anti-lymphoma treatment since randomization, whichever happens first.
Treatment Emergent Adverse Events | 7 Years
  Adverse events reported for the first time or worsening of a pre-existing event after the first dose of study drug/treatment.

IPD SHARING:
Plan to Share IPD: Yes
Incyte shares data with qualified external researchers after a research proposal is submitted. These requests are reviewed and approved by a review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  The trial data availability is according to the criteria and process described on https://www.incyte.com/our-company/compliance-and-transparency
Supporting Information: Study Protocol, SAP
Time Frame: Data will be shared after the primary publication or 2 years after the study has ended for market authorized products and indications.
Access Criteria: Data from eligible studies will be shared with qualified researchers according to the criteria and process described in the Data Sharing section of the www.incyteclinicaltrials.com website. For approved requests, the researchers will be granted access to anonymized data under the terms of a data sharing agreement.
URL: https://www.incyte.com/our-company/compliance-and-transparency